CLINICAL TRIAL: NCT06320704
Title: Occlusal Balance Effect on Mandibular Bone Density by Using Fractal Analysis in Complete Denture Patients (Split-Mouth Study)
Status: Recruiting | Type: Observational
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Shady El Naggar, Associate Professor, Badr University
Other Study IDs: 01067485392
Record Dates: First submitted 2023-05-19; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Bone Density
Keywords: Denture, Fractal, Density

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Complete Denture Group: Completely edentulous patients undergoing complete denture treatment plan effectively balanced using oculosense device
  Interventions: Device: Digital occlusal adjustment using Occulosense digital device

INTERVENTIONS:
Device: Digital occlusal adjustment using Occulosense digital device — Digital occlusal adjustment of mandibular complete denture using Occulosense digital device

SUMMARY:
Although the number of individuals who are edentulous is declining, a sizable fraction still needs a complete denture for their oral rehabilitation.Tooth loss is an issue in public health that determines quality of life since it is linked to socioeconomic, physiological, and psychological aspects. In patients who are completely edentulous, dental implants have been viewed as a favorable choice for rehabilitation.

DETAILED DESCRIPTION:
Although the number of individuals who are edentulous is declining, a sizable fraction still needs a complete denture for their oral rehabilitation.Tooth loss is an issue in public health that determines quality of life since it is linked to socioeconomic, physiological, and psychological aspects. In patients who are completely edentulous, dental implants have been viewed as a favorable choice for rehabilitation.

There have been various occlusion schemes proposed. The term "lingual occlusion," or "LO," was first used in 1941 to describe the occlusion of the mandibular occlusal surfaces with the maxillary lingual cusps in a central and non-centric relationship. This makes it simpler to acquire both the dental position and the occlusal scheme LO.

DeVan suggested the neutral-centric or zero-degree (ZD) occlusion method, in which the cusps are at a zero-degree inclination to balance the incline, centralise the masticatory power, and get around the challenge of attaining precise jaw relations. Moreover, compared to cusped teeth, teeth with a zero-degree occlusal angle exert less pressure on the soft tissues. 13,14 The optimal occlusal scheme in terms of masticatory performance and patient quality of life/satisfaction, however, has not been determined.

Many radiomorphometric studies have employed digital panoramic radiographs to predict osteoporosis based on BMD levels. Dental professionals may employ the mandibular cortical width (MCW), panoramic mandibular index, and Klemetti index as general useful methods to screen for low BMD and anticipate osteoporosis. The meta-analysis determined that the erosion of mandibular cortical bone had an estimated sensitivity and specificity in identifying osteoporosis of 0.806 and 0.643, respectively.

Because individuals with cortical width more than 4 mm typically have normal BMD, MCW also exhibits improved specificity in eliminating osteopenia/osteoporosis. It will be extremely helpful for the initial screening of the osteoporosis risk and advising the assessment of further clinical risk factors to prevent osteoporotic fracture because the panoramic radiograph is frequently employed as a diagnostic tool in dental practice.

Nevertheless, it takes a lot of effort and is prone to measurement errors to manually measure the potential values in a panoramic radiograph. By evaluating the breadth of cortical bone at the mandible, automated osteoporosis detection utilizing digital panoramic radiography is typically carried out to aid doctors. According to a digital panoramic radiograph used in a computer-assisted technique for detecting osteoporosis, there is an about 53% association between cortical bone width and the results of the BMD assessment. In agreement with this, the study by Geary et al. also showed a significant correlation between the width of cortical bone and bone density, though the significance level decreased when other variables, like age, the length and width of the jaw, and the number of teeth, were added to determine bone density.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients ranging from age 45 to 75 years
* Angle's Class I skeletal relationship
* Normal facial symmetry
* Cooperative patients
* Adequate inter-arch space not less than 12mm

Exclusion Criteria:

* Temporomandibular disorders
* Uncontrolled diabetes
* Bleeding disorders or anticoagulant therapy
* Flabby tissues or sharp mandibular residual ridge.
* Heavy smokers.
* Patient's with neuromuscular disorders
* Patients on chemotherapy or radiotherapy
* Severe psychiatric disorders
* Angle's class II and III skeletal relationship

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients present with severe systemic diseases as uncontrolled diabetes, bleeding disorders, neuromuscular disorders, psychiatric disorders and patients on chemotherapy or radiotherapy will be excluded as they will require special management in their drug doses, short appointment visits which will has to be early morning. Furthermore they are more liable to drop out during the follow-up period of the trial.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-03-21 (Estimated); Primary Completion 2024-09-21 (Estimated); Study Completion 2024-09-21 (Estimated)

PRIMARY OUTCOMES:
Bone Density | zero
  Fractal analysis of OPG of mandibular bone
Bone Density | 1 month
  Fractal analysis of OPG of mandibular bone
Bone Density | 3 months
  Fractal analysis of OPG of mandibular bone
Bone Density | 6 months
  Fractal analysis of OPG of mandibular bone

CONTACTS AND LOCATIONS:
Locations (1):
- Badr University in Cairo, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided